CLINICAL TRIAL: NCT03190759
Title: Assessment of the Severity of Acute Asthma Exacerbation in Children Attending the Emergency Departments to Predict Outcomes by Modified Pulmonary Index Score
Brief Title: Assessment of Asthma Exacerbation in Children by Modified Pulmonary Index Score
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hend Heshmat, prinicpal investigator, Assiut University
Other Study IDs: asmpis
Record Dates: First submitted 2017-06-10; First posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Asthma is a heterogeneous disease, usually characterized by chronic airway inflammation. It is defined by the history of respiratory symptoms such as wheeze, shortness of breath, chest tightness and cough that vary over time and in intensity, together with variable expiatory airflow limitation. This definition was reached by consensus, based on consideration of the characteristics that are typical of asthma and that distinguish it from other respiratory conditions .

Asthma is a problem worldwide, with an estimated 300 million affected individuals .It appears that the global prevalence of asthma ranges from 1% to 18% of the population in different countries .

DETAILED DESCRIPTION:
Over the past years, an increase in the number of emergency department (ED) visits for asthma exacerbation has been reported. Most of these visits are for preschool children.

Although pulmonary function tests are commonly used to assess the severity of acute asthma in adults, they are difficult to perform in children, especially those who are younger than five years old .

spirometry measures pulmonary markers such as vital capacity and maximal forced expiatory volume in 1 second. Well-trained personnel are required to perform these tests, and they are not routinely available in the ED. Peak flow has been used in the ED to measure the degree of respiratory obstruction .This technique is difficult to perform in children less than 6 years of age because of their lack of coordination and comprehension .

Adequate evaluation of the severity of asthma exacerbation is important for the initial management of patients, as well as for assessing the clinical response. However, severity is more difficult to assess in children. The clinical evaluation and physician's experience are often not enough to determine the degree of respiratory obstruction .

In the emergency room setting, the most critical issue facing the attending physician is, deciding the adequacy of outpatient therapy of acute asthma, or when hospitalization is indicated. Traditionally, this decision is used to be made according to the clinical history, physical examination, laboratory results and response to therapy of the patient .

A number of asthma severity measures or scoring systems have been established to estimate the degree of airway obstruction for children in whom the standard measurements cannot be performed. These systems combine a number of physical signs, such as respiratory rate and accessory muscle use, to form an aggregate score that estimates the severity of an acute asthma exacerbation .no scoring system is perfect, but some method of assessing severity in children is needed when spirometry testing is not obtainable.

modified the pulmonary index was reported by adding 2 scoring items, namely heart rate and SpO2 at room temperature, and by dividing the method of heart rate and respiratory rate scoring depending on which of 2 age groups the patient belong to. Modified Pulmonary Index Score is a quantitative method of evaluating respiratory conditions in asthmatic subjects modified and consists of 6 evaluation items, which are important for the assessment of dyspnea and are relatively easy to assess in clinical practice, namely heart rate, respiratory rate, accessory muscle use, inspiratory to expiatory flow ratio, degree of wheezing, and oxygen saturation in room air.

the predictive validity and reproducibility of the Modified Pulmonary Index Score for asthma exacerbation was reported in 30 children with a mean age of 7.6 ± 5.5 years in 2005. They found good correlations of the Modified Pulmonary Index Score with clinical outcomes such as ICU admission. The Modified Pulmonary Index Score appears to be suitable for measuring the severity of acute asthma exacerbation, and was applied as primary outcome measurement in some clinical trials .

A significant correlation between Modified Pulmonary Index Score at hospitalization and hospitalization period in children above 5 years old, suggesting that Modified Pulmonary Index Score was useful for predicting the clinical course after hospitalization. However, its applicability to preschool children has not yet been fully elucidated.

The Modified Pulmonary Index Score can be a useful tool for several aspects during acute asthma attacks, including the determination of a treatment plan, and prediction of the period of hospitalization in admitted patients .

ELIGIBILITY:
Inclusion Criteria:

* children with acute asthma exacerbation
* children with acute asthma aged 1-17 years old
* background history of asthma
* this study will deal with the protocols applied in Assiut university children hospital

Exclusion Criteria:.

* children below age of 1 year and more than 17 years old
* Known Tuberculosis exposure
* concurrent stridor
* use of oral corticosteroids in the previous four weeks
* Significant co-morbid disease : lung ,cardiac ,immune , liver , endocrine ,neurological or psychiatric
* children with other causes of respiratory distress
* Children with mild or controlled asthma.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: all patient admitted to emergency department of assiut university within three months of winter of anticipated number 60
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2017-11-11 (Estimated); Primary Completion 2017-12-22 (Estimated); Study Completion 2018-10-20 (Estimated)

PRIMARY OUTCOMES:
ICU admission according to oxygen saturation <81%, respiratory rate <6years old = >60 ≥6years old = >50 and heart rate <3 years old = >160 ≥3 years old= >140 | within 15 minute
  Adequate evaluation of the severity of asthma exacerbation is important for the initial management of patients,using clinical parameters to decide ICU admission :oxygen saturation ,heart rate,respiratory rate and Degree of agitation and conscious level.

SECONDARY OUTCOMES:
hospital stay | within one week
  we will assess all patients with asthma by using parameters which included in modified pulmonary index score"namely heart rate, respiratory rate, accessory muscle use, inspiratory-to expiratory flow ratio, degree of wheezing, and oxygen saturation in room air." using score in predicting hospital stay

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Becker AB, Nelson NA, Simons FE. The pulmonary index. Assessment of a clinical score for asthma. Am J Dis Child. 1984 Jun;138(6):574-6. doi: 10.1001/archpedi.1984.02140440058015. PMID 6720644
- [Result] Gorelick MH, Stevens MW, Schultz TR, Scribano PV. Performance of a novel clinical score, the Pediatric Asthma Severity Score (PASS), in the evaluation of acute asthma. Acad Emerg Med. 2004 Jan;11(1):10-8. doi: 10.1197/j.aem.2003.07.015. PMID 14709423
- [Result] Masoli M, Fabian D, Holt S, Beasley R; Global Initiative for Asthma (GINA) Program. The global burden of asthma: executive summary of the GINA Dissemination Committee report. Allergy. 2004 May;59(5):469-78. doi: 10.1111/j.1398-9995.2004.00526.x. No abstract available. PMID 15080825
- [Result] Smith SR, Baty JD, Hodge D 3rd. Validation of the pulmonary score: an asthma severity score for children. Acad Emerg Med. 2002 Feb;9(2):99-104. doi: 10.1111/j.1553-2712.2002.tb00223.x. PMID 11825832
- [Result] van der Windt D. Promises and pitfalls in the evaluation of pediatric asthma scores. J Pediatr. 2000 Dec;137(6):744-6. doi: 10.1067/mpd.2000.111458. No abstract available. PMID 11113827
- [Result] Weiss KB, Wagener DK. Changing patterns of asthma mortality. Identifying target populations at high risk. JAMA. 1990 Oct 3;264(13):1683-7. PMID 2398607